CLINICAL TRIAL: NCT06331468
Title: Phase II Trial of Hypofractionated Radiochemotherapy for Women With Metastatic or Bulky Uterine Cervix Cancer
Brief Title: Hypofractionated Radiochemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Denise Fabian (Other)
Responsible Party: Sponsor-Investigator, Denise Fabian, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23-GYN-10
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-06

CONDITIONS: Uterine Cervix Cancer
Keywords: Uterine Neoplasm; Cisplatin
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms | interventions — Cisplatin; Radiotherapy, Intensity-Modulated; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cisplatin with concurrent Intensity Modulated Radiotherapy and Brachytherapy (Experimental): Cisplatin two (2) one-time weekly intravenous infusions at 40 mg/m2 (70mg maximum)
  IMRT once daily, four fractions per week for 2 weeks 4.56 Gy x 8 fractions
  High dose rate Brachytherapy twice per week with a 2-day break in between sessions for a total of four brachytherapy treatments. The dose is 7 Gy x 4 fractions
  Interventions: Drug: Cisplatin; Radiation: intensity modulated radiation therapy (IMRT); Radiation: high-dose-rate (HDR) brachytherapy

INTERVENTIONS:
Drug: Cisplatin — A total of two IV infusions of cisplatin will be administered on Day 1 and again on Day 8 +/- 1 day. Cisplatin starting dose is 40 mg/m2. Dose reduction is allowed (30 mg/m2) as needed for management of toxicities.
  Other Names: Platinol
Radiation: intensity modulated radiation therapy (IMRT) — given once daily Monday-Thursday, four fractions per week for 2 weeks. The radiation dose is 4.56 Gy x 8 fractions.
Radiation: high-dose-rate (HDR) brachytherapy — administered 2x weekly (allow at least 72-hours window between sessions); weekdays only for 2 weeks. The radiation dose is 7 Gy x 4 fractions.

SUMMARY:
The goal of this clinical trial is to investigate the use of hypofractionated radiation (delivery of fewer but larger doses of radiation) with concurrent chemotherapy for women with metastatic of bulky uterine cervix cancer. The main questions it aims to answer are:

* What is the MRI-assessed rate of response at 1-month and 3-months post-treatment?
* What is the safety and tolerability of cisplatin-based hypofractionated pelvic Intensity Modulated Radiation Therapy (IMRT) followed by brachytherapy?
* What is the median progression-free survival and overall survival at 1 and 2 years for patients who undergo cisplatin-based hypofractionated pelvic IMRT?
* What is the proportion of patients who complete the treatment in prescribed timeframe?
* What the levels of cervix cancer circulating tumor cells pretherapy and after treatment?

To confirm eligibility, within four weeks prior to study enrollment, all patients will undergo the following:

* Complete history and physical exam, GOG performance status evaluation
* Standard of care scans, which include staging CTs and/or PET scans, and MRI to verify eligibility and appropriate stage of disease. Blood tests will be done to check various organ functions.

Treatment will be administered on an outpatient basis.

The main difference between the proposed regimen in the trial and standard of care is as follows:

1. The trial has a shortened course of EBRT. Standard of care utilizes 25 treatments, also known as "fractions" of EBRT, while the trial utilizes 8 fractions of EBRT. An equivalent "biological effective dose" is achieved by increasing the radiation dose per fraction.
2. The concurrent cisplatin dosing is shortened from 5-6 cycles of cisplatin to 2 cycles of cisplatin. The dose of cisplatin is 40 mg/m2.

This protocol requires photon IMRT technique followed by high dose rate (HDR) brachytherapy. The therapies use focused energy beams to kill cancer cells. Radiation therapy must be completed within 30 days +/- 2 days of initiation. Computed tomography simulation with the patient in a head-first laying on back-supine position is required. MRI-guided treatment planning and image guidance during treatment for motion management will be used.

IMRT will be given once daily Monday-Thursday, four fractions per week. The high-dose-rate (HDR) brachytherapy following institutional protocol. Brachytherapy will be delivered twice per week with a 2-day break in between sessions. A total of four brachytherapy treatments will be delivered.

After active therapy is completed, treatment-related toxicity will be assessed at the 1-month post-treatment completion visit and again at the 3-month post-treatment completion. Patients removed from the study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event(s).

Routine MRI imaging to assess treatment response to radiotherapy is conducted at Day 15. Treatment response to radiotherapy followed by brachytherapy will be assessed at the 1- month and 3-months post-treatment completion.

Following the 3-months post-treatment completion, study participants will be followed for disease progression and survival status until Year 2 post-treatment initiation. NOTE: Cervical cancer patients are routinely followed (clinical surveillance) every 3-months during the first two years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Untreated, pathologically or cytologically-confirmed diagnosis of FIGO Stage IB3, II, or IIIA-IIIC1 bulky ( ≥ 6cm) or Stage IVA or Stage IVB (FIGO 2018) squamous, adenosquamous, or adenocarcinoma of the uterine cervix with limited metastatic burden (not requiring urgent systemic therapy).
* Adequate organ and marrow function
* Gynecologic Oncology Group performance status of 0, 1, or 2
* Patient agrees to use two forms of birth control if they are of child-bearing potential
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Presence of another concurrent active invasive malignancy
* Prior invasive malignancy diagnosed within the last three years, with the following two exceptions: [a] non-melanoma skin cancer and/or [b] prior in situ carcinoma of the cervix
* Receipt of prior pelvic radiotherapy for any reason that would contribute radiation dose that would exceed tolerance of normal tissues, at the discretion of the treating physician
* Currently receiving any other investigational agent(s) for the treatment of cancer
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Cisplatin or other agents used in study
* Presence of uncontrolled intercurrent illness as determined by the treating physician
* pregnant or lactating
* Patients with a known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
MRI assessed rate of complete response | 1 month post treatment (day 60)
  MRI-assessed rates of complete response as estimated by the number of CRs (complete response per RECIST v1.1) divided by the total number of evaluable subjects

SECONDARY OUTCOMES:
MRI assessed rate of complete response | 3 months post treatment (day 120)
  The proportion of complete response will be assessed at 3-mos post-treatment completion, i.e., Day 120, as estimated by the number of CRs (complete response per RECIST v1.1) divided by the total number of evaluable subjects.
progression-free survival (PFS) | up to 2 years
  Progression-free survival (PFS) is calculated from the date of treatment start (week 1, day 1) to the date of initial disease progression or to the date of death or to 2-years post-treatment initiation, whichever occurs first.
overall survival (OS) | up to 2 years
  Overall Survival is calculated from the date of treatment start until date of death or up to 2-years post-treatment initiation, whichever occurs first.
Treatment Completion | up to 32 days
  reported as a proportion of subjects who complete entire prescribed course of the treatment based on the treatment compliance for Radiotherapy and for Cisplatin
Treatment Tolerability | up to 2 years
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE v4.0)

OTHER OUTCOMES:
Change in levels of uterine cervix cancer circulating tumor cells | pre-treatment; 1-month post-treatment completion (Day 60); and 3-mos post-treatment completion (Day 120)
  A total of 15mL of peripheral venous blood will be collected for Circulating tumor cells (CTC). Counts will be reported as means with standard deviations in tabular format

CONTACTS AND LOCATIONS:
Overall Officials: Denise Fabian, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No